CLINICAL TRIAL: NCT04736914
Title: A Perspective Study of Zanubrutinib-based Induction and Maintenance Therapy in Young and Fit Patients With Untreated Mantle Cell Lymphoma (BRIDGE)
Brief Title: Zanubrutinib-based Induction and Maintenance Therapy in Young and Fit Patients With Untreated Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huiqiang Huang, Chief Physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-2002-IIT
Record Dates: First submitted 2021-02-01; First posted 2021-02-03 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Intervention Model Description: Zanubrutinib Combined with R-CHOP，R-DHAOx
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zanubrutinib+R-CHOP/R-DHAOx (Experimental): Induction:
  Alternating 3× R-CHOP/ 3× R-DHAOx, every 21 days plus oral Zanubrutinib in cycle 1, 3, 5 in combination with R-CHOP:
  ASCT conditioning
  Maintenance:
  * Zanubrutinib, 160mg PO BID, continuously for 2 year
  * Zanubrutinib maintenance will start after regeneration of peripheral blood count after the end of the last cycle of induction therapy or ASCT
  Requirements for start of maintenance:
  * ANC ≥ 1,000 cells/mm³ (1.0 X 109/L);
  * Platelets ≥ 50,000 cells/mm³ (50 X 109/L);
  Interventions: Drug: R-CHOP/R-DHAOx； Zanubrutib（induction）； ASCT conditioning ； Zanubrutinib（Maintenance）

INTERVENTIONS:
Drug: R-CHOP/R-DHAOx； Zanubrutib（induction）； ASCT conditioning ； Zanubrutinib（Maintenance） — Alternating 3× R-CHOP/ 3× R-DHAOx, every 21 days plus oral Zanubrutinib in cycle 1, 3, 5 in combination with R-CHOP:
  R-CHOP (cycle 1,3,5):
  Rituximab 375 mg/m2 D1, I.V. Cyclophosphamide 750 mg/m2 D1, I.V. Doxorubicine 50 mg/m2 D1, I.V. Vincristine 1.4mg/m2(max 2mg)D1, I.V. Prednisone 100mg D1-5, oral Zanubrutinib 160mg BID D1-21, oral
  R-DHAOx (cycle 2,4,6):
  Dexamethasone 40mg D1-4 oral/I.V. Rituximab 375mg/m2 D1, I.V. Ara-C 2×2g/m2 q12h D2, I.V. Cisplatin 100mg/m2 D1, I.V.
  Maintenance:
  * Zanubrutinib, 160mg PO BID, continuously for 2 year or until progressive disease。
  * Zanubrutinib maintenance will start after regeneration of peripheral blood count after the end of the last cycle of induction therapy or ASCT
  Other Names: R-CHOP，R-DHAOx，Brukinsa

SUMMARY:
This is a prospective, single-center, single-arm, phase II study of Zanubrutinib-based induction followed by ASCT and Zanubrutinib maintenance (2 years) or followed directly by Zanubrutinib maintenance without ASCT in young and fit patients with untreated MCL.

There will be an initial safety run-in phase of 6 patients which will be closely monitored for the observed toxicities during cycle1 in， induction therapy. After completion of safety run-in phase, the investigator will assessed and decided whether to continue the trial as planned. If no unexpected toxicity has been observed, study will expand the sample size to further assess efficacy and safety.

Total around 47 patients aged 18-65 years with previously untreated, Ann Arbor stage II-IV, histologically proven MCL will be enrolled to receive alternating 3 cycles R-CHOP + Zanubrutinib /3 cycles R-DHAOx induction. Totally 6 cycles in induction and every 21 days per cycle. Due to lack of published data about BTKi in combination with R-DHAOx, Zanubrutinib is only applied in cycle 1,3,5(R-CHOP), 160mg BID, d1-21, and not in combination with R-DHAOx

Patients who achieve remission (≥PR) will be allowed to proceed to ASCT or maintenance. Whether ASCT or not depends on investigator's evaluation and discretion. In patients who do not achieve a remission at end of induction (treatment failure), no study specific treatment is defined; rather, the further salvage treatment is upon the discretion of investigators. Patients remain in study for progression and survival follow-up.

Patients will receive Zanubrutinib maintenance for two years in case of remission at ASCT assessment or end of induction assessment. Zanubrutinib is applied oral 160mg BID, continuously for 2 year or until progressive disease, unacceptable toxicity or death, whichever comes first.

The primary analysis will be performed after last-patient completes induction treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Histologically confirmed diagnosis of MCL according to WHO classification
2. Previously untreated MCL
3. Suitable for high-dose treatment including high-dose Ara-C
4. Age ≥ 18 years and ≤ 65 years
5. Stage II-IV (Ann Arbor)
6. Measurable disease by computed tomography (CT)/magnetic resonance imaging (MRI). Measurable disease was defined as at least 1 lymph node > 1.5 cm in longest diameter and measurable in 2 perpendicular dimensions; in case of bone marrow infiltration only, bone marrow aspiration and biopsy are mandatory for all staging evaluations
7. ECOG performance status ≤ 2
8. The following laboratory values at screening (unless related to MCL):

   * Absolute neutrophil count (ANC) ≥ 1×10⁹/L
   * Platelets ≥ 75×10⁹/L (platelets ≥ 50×10⁹/L with bone marrow involvement)
   * Transaminases (AST and ALT) ≤ 3 × upper limit of normal (ULN)
   * Total bilirubin ≤ 2 × ULN (unless documented Gilbert's syndrome)
   * Calculated creatinine clearance ≥ 30 mL/min
9. International normalized ratio ≤ 1.5 and activated partial thromboplastin time ≤ 1.5 x upper limit of normal. If a factor inhibitor was present with prolongation of the international normalized ratio or activated partial thromboplastin time.
10. Sexually active men and women of child-bearing potential must agree to use highly effective contraceptives (eg, condoms, implants, injectables, combined oral contraceptives, intrauterine devices, sexual abstinence, or sterilized partner) while on study; this should be maintained for 90 days after the last dose of study drug
11. Life expectancy of> 3 months
12. Written informed consent form according to GCP and national regulations

Exclusion Criteria:

1. Known CNS involvement of MCL
2. Major surgery within 4 weeks of screening
3. Prior hematopoietic stem cell transplantation
4. Concomitant or previous malignancies within the last 2 years other than basal cell skin cancer or in situ uterine cervix cancer
5. Clinically significant cardiovascular disease such as uncontrolled arrhythmias and hypertension , congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification or LVEF below 50%（AHA，2016）
6. QTcF > 450 msec or other significant electrocardiogram (ECG) abnormalities including second-degree atrioventricular block Type II, or third-degree atrioventricular block
7. Clinically significant hypersensitivity (eg, anaphylactic or anaphylactoid reactions to the compound of zanubrutinib itself or to the excipients in its formulation)
8. Requires treatment with strong CYP3A inhibitors or strong CYP3A inducers
9. Unable to swallow capsules or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
10. Patients with unresolved hepatitis B or C infection or known HIV positive infection
11. Active infection including infections requiring oral or intravenous antimicrobial therapy
12. Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could have compromised the patient's safety, or put the study at risk
13. History of stroke or intracranial hemorrhage within 6 months before first dose of study drug
14. Pregnancy or lactation
15. Participation in another clinical trial within 30 days before enrollment in this study
16. poor compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2021-01-31 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
MRD negativity rate | 18 weeks
  To evaluate the MRD negativity rate after Zanubrutinib-based induction therapy in subjects with newly diagnosed, young and fit MCL.
  The primary endpoint of the trial will be bone marrow minimal residual disease (MRD) negative rate after induction therapy (at the completion of cycle 6 or at premature discontinuation).

SECONDARY OUTCOMES:
Duration of MRD negativity | 60 months
  The time from the first achieving MRD negativity after start of treatment to the MRD convert to positive
Progression free survival (PFS) | 60 months
  The time from start of treatment to progression or death from any cause
Overall survival (OS) | 60 months
  The time from start of treatment to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No